CLINICAL TRIAL: NCT03247647
Title: Enhancing the Efficacy and Duration of a Brief Alcohol Intervention Using Self-Affirmation
Brief Title: Personal Values and Mandated Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Binghamton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1708001882; 1R01AA025643-01 (NIH)
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Abuse
Keywords: Alcohol Intervention; College Students
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Intervention (Experimental): Participants assigned to this arm will complete a personal values task before reviewing their personalized feedback (eCheckUpToGo).
  Interventions: Behavioral: Enhanced Intervention
- Standard Intervention (Placebo Comparator): Participants assigned to this arm will complete a writing task about the food they have eaten in the past 48 hours immediately before reviewing their personalized feedback (eCheckUpToGo).
  Interventions: Behavioral: Standard Intervention

INTERVENTIONS:
Behavioral: Enhanced Intervention — Participants will complete a personal values task immediately before viewing feedback from eCheckUpToGo.
  Arms: Enhanced Intervention
Behavioral: Standard Intervention — Participants will write about the food they have eaten in the last 48 hours.
  Arms: Standard Intervention

SUMMARY:
This study aims to examine the efficacy of an enhanced alcohol intervention among individuals who are mandated to complete an alcohol education activity as part of a university sanction.

DETAILED DESCRIPTION:
High volume drinking and related adverse consequences pose significant health concerns at US colleges and universities; drinking behavior often leads to students being sanctioned for violations of campus alcohol policy. Given the widespread use of mandated alcohol interventions for these students, optimizing their initial effects and their duration could substantially mitigate adverse alcohol outcomes. Self-affirmation represents a promising adjunct to brief alcohol interventions, particularly those delivered via computer that are popular but tend to have smaller effects. Basic research shows that when self-affirmation exercises precede the receipt of health information, they decrease defensiveness and resistance to threatening health information and increase acceptance and processing of health messages. Furthermore, the facilitative effects of self-affirmation are strongest among those at higher risk. Because many mandated students display both defensiveness and high drinking severity, use of self-affirmation to enhance information processing and reduce defensive responding could optimize the efficacy of an active alcohol intervention in this at-risk subpopulation. The investigators propose to use a two-group randomized design to investigate the effect of a self-affirmation exercise prior to an empirically supported brief alcohol intervention consisting of computer-delivered personalized normative feedback (PNF). Building on an extensive history of academic-student affairs collaborations, the investigators will recruit 450 mandated students from a large public university over the course of 5 semesters. The primary aim is to examine the additive effects of an initial self-affirmation (SA) manipulation prior to receiving PNF (SA + PNF) relative to Control + PNF on alcohol use and consequences. This study extends prior work by evaluating the ability of self-affirmation exercises to supplement active alcohol interventions (rather than just health messages), and tracking the impact on alcohol use over a longer (12-month) follow-up period. Secondary aims include (a) testing theoretically-derived mediation sequences that explain the SA + PNF effects on alcohol use and alcohol consequences, incorporating mechanisms of action associated with both self-affirmation and brief alcohol interventions, and (b) the examination of theoretical moderators of the effects of SA + PNF on alcohol use and alcohol consequences. The investigators will use latent growth curve modeling analyses to examine direct and indirect intervention effects on alcohol use and consequence trajectories from (pre-intervention) baseline assessment across 1-, 3-, 6-, 9- and 12-month follow-ups. The public health goal of this research is to reduce the acute and chronic effects of alcohol misuse by improving the efficacy of a low intensity brief alcohol intervention. The findings of this study have both practical and theoretical implications. Demonstration of the additive utility of a very brief self-affirmation exercise could improve the efficacy and impact of currently available computer-delivered interventions for mandated students; it may also expand the reach of self-affirmation theory, leading to adaptation of self-affirmation for use with other at-risk populations receiving brief alcohol interventions.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years of age
* Enrolled in the university's undergraduate four-year degree program
* Have been mandated for violation of university alcohol policy.

Exclusion Criteria:

- Seniors who will graduate before the final 12-month follow-up

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 486 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Alcohol Consumption | 1 month after baseline
  Average of reports from past 30 days on the number of standard drinks consumed by participant per week.

SECONDARY OUTCOMES:
Alcohol-related consequences | 1 month and 3 months after baseline
  Participant self-report on the Brief Young Adult Alcohol Consequences Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kate B Carey, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Binghamton University, Binghamton, New York
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and the results of the study have been published, de-identified data will be made available to other qualified investigators upon request. The request will be evaluated by the investigators to ensure that it meets reasonable demands of scientific integrity.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Within one year of study completion
Access Criteria: To be determined

REFERENCES:
- [Derived] Carey KB, DiBello AM, Magill M, Mastroleo NR. Does self-affirmation augment the effects of a mandated personalized feedback intervention? A randomized controlled trial with heavy drinking college students. Psychol Addict Behav. 2024 Dec;38(8):836-849. doi: 10.1037/adb0000989. Epub 2024 Jan 18. PMID 38236233
- [Derived] Hatch MR, Wilson SE, Mastroleo NR, DiBello AM, Carey KB. Values of College Students Mandated to an Alcohol Intervention: A Qualitative Examination. Subst Use Misuse. 2022;57(14):2094-2100. doi: 10.1080/10826084.2022.2136492. Epub 2022 Oct 31. PMID 36315498
- [Derived] Wilson SE, Feltus SR, Brenman AM, Carey KB, DiBello AM, Mastroleo NR. Comparing Alcohol Use of Pre-COVID-Era and COVID-Era Cohorts of Mandated College Student Drinkers. J Stud Alcohol Drugs. 2022 Jul;83(4):480-485. doi: 10.15288/jsad.2022.83.480. PMID 35838424